CLINICAL TRIAL: NCT04849754
Title: Analysis of the Evolution of SUVmax by Quantitative Analysis Method of Bisphosphonate Scintigraphy for the Follow-up of Patients With Transthyretin Amyloidosis Treated With Tafamidis
Brief Title: Analysis of the Evolution of SUVmax by Quantitative Analysis Method of Bisphosphonate Scintigraphy
Acronym: QUANTI-SUV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A01795-34
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with transthyretin related cardiac amyloidosis (Other): Bone scintigraphy
  Interventions: Diagnostic Test: bone scintigraphy

INTERVENTIONS:
Diagnostic Test: bone scintigraphy — Bone scintigraphy

SUMMARY:
Recently, treatment with tafamidis in patients with cardiac ATTR lead to a significant reduction in mortality. The Perugini score is commonly used on planar bone scans to differentiate cardiac ATTR from other amyloidosis or normal patients but fails to evaluate amyloid burden and patient prognosis. Although semi-quantitative methods have been suggested to evaluate the amyloid burden, there a need for quantitative methods for longitudinal assessment of the disease.

DETAILED DESCRIPTION:
Cardiac amyloidosis is a cause of restrictive cardiomyopathy with preserved ejection fraction associated with amyloid fibrils deposits in the myocardium. Two types of amyloid commonly infiltrate the heart: immunoglobulin light-chain amyloid (AL), and transthyretin-related amyloid amyloidosis (ATTR). Cardiac imaging is currently used for the diagnosis of ATTR, including planar scintigraphy with bone seeking radiopharmaceuticals, cardiac magnetic resonance and echocardiography with global longitudinal strain assessment.Although semi-quantitative methods have been suggested to evaluate the amyloid burden, there a need for quantitative methods for longitudinal assessment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age
* Patient diagnosed with transthyretin cardiac amyloidosis confirmed by scintigraphy
* Patient with signed consent

Exclusion Criteria:

* Patients with systemic AL amyloidosis
* Protected patient : major under guardianship, tutorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of SUVmax by quantitative analysis by bisphosphonate scintigraphy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fredric MOUQUET, Principal Investigator — Hôpital Privé Le Bois
Locations (1):
- Hôpital privé Le Bois, Lille, France

IPD SHARING:
Plan to Share IPD: No